CLINICAL TRIAL: NCT06454162
Title: Effect of Adding Modified Ketogenic Diet to Exercise Program in Treating Obese Patient With Multiple Sclerosis: A Randomized Controlled Trial
Acronym: MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator nabil mahmoud ismail abdel-aal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005184
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
Keywords: Modified Ketogenic Diet; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Modified Ketogenic Diet and exercise program
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Ketogenic Diet (Experimental): thirty-two patients will receive modified ketogenic diet and exercise program for three months
  Interventions: Other: Modified Ketogenic Diet; Other: exercise program
- exercise program (Active Comparator): thirty-two patients will receive an exercise program three times per week for three months
  Interventions: Other: exercise program

INTERVENTIONS:
Other: Modified Ketogenic Diet — the patients will receive KD after nutritional counseling, patients will instructed to start by limiting carbohydrate intake to just 20 g/day for 4 weeks in order to establish ketosis. Then, patients increase their carbohydrate intake by 5 g each week until they reach their individual maximum (approximately 40 g) to maintain stable ketosis. All carbohydrates relevant for elevating blood glucose are limited to 40-50 g/ day. In addition, the glycemic index and glycemic load of carbohydrates have to be below 50 and 60, respectively. This ketogenic diet is equivalent to a traditional ketogenic diet, but with a liberalized macronutrient composition of 70-80% fats, 15-20% proteins and 5-10% carbohydrates (compared to a traditional ketogenic diet with 90% fat, 6% proteins and 4% carbohydrates)+ exercise program
  Arms: Modified Ketogenic Diet
Other: exercise program — the patients will receive exercise program in the form of aerobic training (10-30 minutes at moderate intensity) and resistance training (1-3 sets of 8-15 repetition maximum (RM)

SUMMARY:
this study will be conducted to investigate the effect of adding Modified Ketogenic diet to exercise program in treating obese patient with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the most common inflammatory disease of the central nervous system in young adults that may lead to progressive disability. Since pharmacological treatments may have substantial side effects, there is a need for complementary treatment options such as specific dietary approaches. Ketone bodies that are produced during fasting diets (FDs) and ketogenic diets (KDs) are an alternative and presumably more efficient energy source for the brain.Ketogenic diets (KDs) are high-fat, low-carbohydrate diets that mimic a fasting state. KDs create a metabolic shift from glycolytic energy production toward oxidative phosphorylation energetics by using fatty acids as a primary source of energy. As these fatty acids undergo beta-oxidation, ketones are produced. This increase in oxidative phosphorylation coupled with ketone production modifies the tri carboxylic acid cycle to limit reactive oxygen species generation. In addition, ketone bodies transported across the blood-brain barrier up regulate antioxidant pathway genes (particularly via the Nrf2 pathway) and boost energy production in brain tissue.sixty-four subjects with MS, ranged from 18-50 years. will be selected randomly divided into two groups each group consists of thirty-two subjects; experimental group (modified ketogenic diet+ aerobic exercise) and control group (aerobic exercise).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS based on McDonald Criteria.
* Patients had to be fully ambulatory, not requiring assistive devices.
* The ages of 18 and 50
* Patients Body mass index (BMI) less than 30 Kg/m2.

Exclusion Criteria:

* Evidence of active disease or relapse phase within the last 30 days
* Chronic heart failure, cancer, chronic kidney disease, infection with human Immunodeficiency
* Addiction to drugs or alcohol.
* Pregnancy and Diabetic patient.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
VO2 max | up to three months
  VO2 max will be measured by cardiopulmonary exercise testing. Maximum level of oxygen consumption definite indicator of muscular work capacity Normal Range = 1,700 - 5,800 ml / min

SECONDARY OUTCOMES:
exercise capacity | up to three months
  six minute walk test will be used to assess the exercise capacity.
fatigue | up to three months
  Modified Fatigue Impact Scale will be used to assess fatigue. participants rate on a 5-point Likert scale, with 0 = 'Never' to 4 = 'Almost always' their agreement with 21 statements. Total score (0-84) and subscales for physical (0-36), cognitive (0-40) and psychosocial functioning (0-8).
life disability | up to three months
  Multiple sclerosis quality of life questionnaire will be used to assess life disability. MSQoL-54 scale scores were created using the Likert method by averaging items within the scales and, then row scores were linearly transformed into 0-100 scales. Higher values indicate better quality of life.
Oxygen Consumption | up to three months
  Oxygen Consumption will be measured by cardiopulmonary exercise testing. Normal = 250 ml / min 3.5 - 4 ml / min / kg, increases directly with the level of muscular work increases until exhaustion occurs and until individual reaches
Carbon Dioxide Production | up to three months
  Carbon Dioxide Production will be assessed by cardiopulmonary exercise testing.Normal = 200 ml / min 2.8 ml / min / kg At Exercise: initial phase, increases at same rate as VO2, once Anaerobic Threshold (AT) is reached, increases at a faster rate than VO2; increase is due to increased acid production I
Anaerobic Threshold | up to three months
  Anaerobic Threshold will be measured by cardiopulmonary exercise testing.Normal: occurs at about 60% of VO2 max, followed by breathlessness, burning sensation begins in working muscles.
Ventilatory Equivalent for Carbon Dioxide | up to three months
  Ventilatory Equivalent for Carbon Dioxide will be measured by cardiopulmonary exercise testing.Minute ventilation / VCO2, to estimate Efficiency of ventilation and Liters of ventilation to eliminate 1 L of CO2.
Ventilatory Equivalent for Oxygen | up to three months
  Ventilatory Equivalent for Oxygen will be measured by cardiopulmonary exercise test. Minute ventilation / VO2, indicate Liters of ventilation per L of oxygen